CLINICAL TRIAL: NCT00377000
Title: A Pilot, Multi-Center, Patient Preference Study Comparing Two Clindamycin/Benzoyl Peroxide Gels.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DL6021-0505
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide

INTERVENTIONS:
Drug: clindamycin 1% / benzoyl peroxide 5% gel pump
Drug: clindamycin 1% / benzoyl peroxide 5% tube

SUMMARY:
Evaluate patient preference factors comparing two clindamycin/benzoyl peroxide gels. One dispensed in a pump presentation, the other in a tube presentation.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

INCLUSION CRITERIA:

1. Patients with a clinical diagnosis of acne vulgaris of mild to moderate severity
2. Females of childbearing potential, in addition to having a negative urine pregnancy test at Visit 1, must be willing to use an acceptable form of birth control during the study.
3. Patients 18 years of age or older must provide Institutional Review Board (IRB) approved written informed consent. Patients under 18 years of age must have IRB approved written informed consent from a parent or legal guardian. Patients 12 - 17 years of age must complete an IRB approved assent form for minors.
4. Patients must be willing and able to understand the requirements of the study, abide by the restrictions, apply the medication as instructed, and return for the required study visits.
5. Patients must be in good health and free from any clinically significant disease, other than acne vulgaris, that might interfere with the study evaluations.
6. Patients who use make-up must have used the same brand of make-up for a minimum period of 2 weeks prior to Baseline and agree to not change make-up brands or types during the study.

EXCLUSION CRITERIA:

1. Patients who are pregnant, nursing, or planning a pregnancy within the study period.
2. Patients who have more than 2 nodulo-cystic lesions on the face, excluding the nose.
3. Patients who have a known hypersensitivity to any ingredients in the test products including clindamycin and benzoyl peroxide.
4. Patients who have been treated with prescription and/or over-the-counter topical products, or had a procedure performed that may impact study assessments.
5. Patients who have any systemic or dermatological disorder that has the potential to interfere with the evaluations (e.g., rosacea, seborrheic dermatitis, perioral dermatitis, corticosteroid-induced acne vulgaris, carcinoid syndrome, mastocytosis, acneform eruptions caused by medication, facial psoriasis, facial eczema, etc.).
6. Patients with clinically significant unstable medical disorders, life-threatening disease, or current malignancies.
7. Patients who engage in activities that involve excessive or prolonged exposure to sunlight.
8. Patients who consume excessive amounts of alcohol, abuse drugs, or have any condition that would compromise compliance with this protocol.
9. Patients who have been treated with an investigational drug or investigational device within a period of 30 days prior to study entry.
10. Alcoholic toners, astringents, medicated topical preparations (prescriptions and over-the-counter), or medicated make-up on the facial treatment area.
11. Abrasive cleansers or washes to the facial area.
12. New cosmetics, or new cleansers applied to the face.
13. Patients must not wear make-up at the visits, so as not to interfere with the evaluations.
14. Patients should not use a sauna within 48 hours prior to each visit.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2005-11; Study Completion 2006-03

PRIMARY OUTCOMES:
Patient Preference Questionnaire evaluation: including product use, patient knowledge and impression of acne, as well as patient treatment
The incidence of all adverse events reported during the study will be summarized by treatment group
The signs and symptoms of irritation will be summarized descriptively by treatment group at every visit
Investigator irritation grading - erythema, peeling, dryness and pruritus at Baseline (Week 0), Week 2, 4, and 6

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, MT, ASCP, Study Director — Sanofi